CLINICAL TRIAL: NCT00991731
Title: A Faith-Based Intervention to Increase Physical Activity Among Blacks
Brief Title: A Program to Increase Physical Activity Among Blacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melicia Whitt-Glover (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Montana State University (Other); Kaiser Permanente (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Melicia Whitt-Glover, President & CEO, Gramercy Research Group
Organization: Gramercy Research Group (Other)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: REE1-09-063; 1R01HL094580-01A1 (NIH)
Record Dates: First submitted 2009-10-06; First posted 2009-10-08 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Physical Activity
Keywords: Physical Activity; Faith based; Non faith based; African American; Female; Pedometers
MeSH Terms: conditions — Motor Activity | interventions — Faith-Based Organizations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Faith-based (Active Comparator): Faith-based interventions incorporate tenets of the faith-based organization (e.g., religious beliefs, scriptural references) and involve the faith-based organization in the planning of the intervention from beginning to end
  Interventions: Behavioral: Faith-based
- Non-faith-based (Active Comparator): A curriculum designed for delivery without biblical references. In the traditional teachings of how to increase physical activity.
  Interventions: Behavioral: Non-faith-based
- Control (No Intervention): This group will receive a printed pamphlet "Energize Yourself! Stay Physically Active", published by the National Heart Lung and Blood Institute, that encourages participation in at least 30 minutes of daily physical activity all at once or in bouts lasting 10 minutes at a time.

INTERVENTIONS:
Behavioral: Faith-based — The faith-based intervention will include 24 group sessions. Sessions 1 - 16 will occur weekly, sessions 17 - 20 will occur bi-weekly, and sessions 21 - 24 will occur monthly. Sessions will be scheduled to last for 90 minutes each. This will include a 30-minute physical activity session (led by a trained exercise leader) and 60 minutes of group discussion (led by a Community Health Worker trained in group facilitation, familiarity with theology and health ministry education, and experience implementing group-based activities in faith settings). Group discussion content will be standardized to ensure consistent delivery. All items will be delivered with biblical references to further guide the participants.
  Arms: Faith-based
Behavioral: Non-faith-based — The non-faith based intervention will include 24 group sessions. Sessions 1 - 16 will occur weekly, sessions 17 - 20 will occur bi-weekly, and sessions 21 - 24 will occur monthly. Sessions will be scheduled to last for 90 minutes each. This will include a 30-minute physical activity session (led by a trained exercise leader) and 60 minutes of group discussion (led by a Community Health Worker trained in group facilitation, familiarity with theology and health ministry education, and experience implementing group-based activities in faith settings). Group discussion content will be standardized to ensure consistent delivery. All items will be delivered without biblical references as in the faith-based intervention.
  Arms: Non-faith-based

SUMMARY:
The purpose of this research study is to evaluate three different approaches for increasing physical activity in African American women who are not currently doing enough physical activity. One approach will teach people about physical activity, in groups, using general principles (general physical activity program). The second approach will teach people about physical activity, in groups, using principles from the bible (faith-based physical activity program). The third approach will teach people about physical activity by giving them written materials created at the National Institutes of Health (control group). Control groups are used in research studies to see if the program being studied really does have an effect on physical activity. At the end of the study, people in the control group will also participate in either the general physical activity program or the faith-based physical activity program.

DETAILED DESCRIPTION:
The intervention will be conducted in 24 churches. Participating churches will be recruited from the list of churches that participated in the Health Ministry Institute, a program including ~40 minority-serving churches in Forsyth County conducted by Dr. Whitt-Glover 2 years ago. We will enroll churches from the list of participating HMI churches over a two-year period until 24 churches have been recruited for randomization. If we exhaust the list of HMI before we have 24 churches enrolled in the study, we will place advertisements in local newspapers and send out directed mailings to the ~210 minority-serving churches in Forsyth County, NC explaining the study and inviting them to send a representative to a study information session to learn more.

Eligible participants will include 480 African American women > 18 years of age who report that they are not currently meeting the guidelines for regular moderate or vigorous physical activity. Participants should have no physical limitations or disabilities that would limit physical activity participation. In addition, participants should have no contraindications for increasing daily physical activity, such as recent myocardial infarction or congestive heart failure, and should be willing to participate in a two-year study.

Participants in the active intervention will participate in 24 group sessions. Sessions 1 - 16 will occur weekly, sessions 17 - 20 will occur bi-weekly, and sessions 21 - 24 will occur monthly. Sessions will be scheduled to last for 90 minutes each. This will include a 30-minute physical activity session (led by a trained exercise leader) and 60 minutes of group discussion (led by a Community Health Worker trained in group facilitation, familiarity with theology and health ministry education, and experience implementing group-based activities in faith settings). Group discussion content will be standardized to ensure consistent delivery.

Thirty-Minute Physical Activity Session. At the beginning of each weekly meeting and immediately prior to the group discussion, participants will engage in a standard 30-minute physical activity session led by a trained exercise leader. The 30-minute physical activity session will include warm-up, an activity period, and cool down. Inclusion of an exercise period during the weekly sessions proved to be a motivator for on-time arrival to weekly sessions during the pilot study, as well as an opportunity for participants to learn methods for proper warm-up and cool-down prior to and following physical activity, as well as time to rehearse using physical activity incentives (e.g., exercise tapes, hand weights), and to understand the body's physiological reactions to moderate-intensity physical activity (i.e., many participants in the pilot study were not exactly sure what moderate-intensity physical activity felt like (e.g., how hard should they be breathing, what should heart rate be?) and may not have engaged in the appropriate intensity-level for physical activity outside of class without opportunities to rehearse activity in class).

Group-Based Intervention Sessions. The group discussion sessions will be led by a Community Health Worker and the format will be similar for each group and will include five segments:

1. Prayer/scripture and check-in (5 minutes). To ensure the cultural appropriateness of the intervention each session in both active arms of the intervention will begin with prayer and reading of an assigned scripture, and will end with prayer, as most church-based activities begin and end this way. By deliberately writing this into both the faith-based and non-faith-based intervention, we can control the amount of spirituality that will be naturally incorporated into the non-faith-based curriculum, which has been a limitation in previous studies comparing faith- and non-faith-based curricula.
2. Review of participant progress in implementing the strategies recommended for changing their physical activity in the previous session (10 minutes). We will use the five-step approach from the continuous care problem-solving model for this segment. The underlying assumption is that problems are a normal part of behavior change and that solutions must be tailored to each individual. The 5 steps include: 1) problem orientation, 2) problem definition and formulation, 3) generation of alternatives, 4) systematic decision making, and 5) implementation and verification. The group leaders will encourage participants to openly describe the progress they have achieved, and to identify any problems they might have encountered. Good progress will be highlighted with strong positive feedback. Difficulties will be dealt with through group support and advice.
3. Skill training (30 minutes) will be related to the new content to be presented during the session and cognitive-behavioral self-management skills (e.g., goal setting, self-monitoring). Content will be delivered from a faith-based perspective incorporating biblical principles or from a non-faith-based perspective that does not include biblical principles.
4. Goal setting (10 minutes). Participant will be asked to identify specific behavioral goals for the next period and will receive feedback and encouragement from the group.

Participants will be compensated for completing all three rounds of data collection. Participants who miss a scheduled data collection visit will be contacted for up to two weeks after the missed visit to attempt to collect the data. At minimum, participants will be asked to report pedometer steps to ensure collection of data related to the primary variables of interest.

Pedometer-Assessed Daily Walking. Daily walking will be measured using a pedometer and a physical activity log in which to record the daily number of steps taken by each study participant. Studies have demonstrated the feasibility of the pedometer both as an objective measure of physical activity and as a potential motivator to increase physical activity levels. All participants will receive the New Lifestyle Pedometer 2000 (NL-2000) at the beginning of the study, and will be asked to keep a record of daily walking on a study log sheet throughout the active intervention period. The NL-2000 also stores walking data for up to 7 days and automatically resets at the beginning of each day, reducing participant burden to remember to reset and record pedometer data each day, and also increasing the likelihood that we will be able to collect complete data on walking for all participants. Participant logs will be reviewed, and feedback will be provided, at the beginning of each group session during the review of participant progress. Participants will measure walking using the NL-2000 daily throughout the active intervention phase.

Accelerometer-Assessed Daily Moderate-to-Vigorous Physical Activity. Participation in daily bouts of moderate-to-vigorous physical activity will be assessed using the Actical Accelerometer (MiniMitter Company, Inc, Bend, OR). Participants will wear wrist-mounted accelerometers for seven consecutive days (one week) at the baseline, 10 month, and 22 month data collection visits. Several continuous variables may be calculated from accelerometer data, including total daily energy expenditure through physical activity, total daily participation in inactivity and light-, moderate-, and vigorous-intensity activity, the average length of each bout of activity at a given intensity level, adherence to the moderate- and vigorous-intensity physical activity recommendations, and adherence to the recommended bout length.

Self-efficacy will be assessed as self-regulatory efficacy and performance efficacy. A barriers self-efficacy scale will be employed as a means of evaluating a key self-regulation process component of the social cognitive framework for the intervention, that is, problem solving necessary to address barriers in their pursuit of changing lifestyle behaviors. The physical activity measure is a 14-item scale that is predictive of 6-month and 1-year adherence to physical activity.

ELIGIBILITY:
Inclusion Criteria:

* African American women > 18 years of age who report that they are not currently meeting the guidelines for regular moderate or vigorous physical activity.
* No physical limitations or disabilities that would limit physical activity participation.
* No contraindications for increasing daily physical activity, such as recent myocardial infarction or congestive heart failure, and should be willing to participate in a two-year study.

Exclusion Criteria:

* Individuals <18 years of age will be ineligible for participation.
* Those with walking aids (e.g., walkers, canes).
* Those who may need additional medical clearance (e.g., severe obesity) will be asked to obtain clearance prior to formal enrollment into the study.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2009-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Comparing the efficacy of faith-based vs non-faith-based to a control condition in increasing daily physical activity measured as steps/day. | baseline, 10 months, and 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Melicia C Whitt-Glover, Ph.D., Principal Investigator — Gramercy Research Group
Locations (1):
- Gramercy Research Group, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Story CR, Gross TT, Harvey IS, Whitt-Glover MC. Pastoral perceptions of the learning and developing individual exercise skills (L.A.D.I.E.S.) intervention: a qualitative study. Health Educ Res. 2017 Feb 1;32(1):81-95. doi: 10.1093/her/cyw054. PMID 28052931
- [Derived] Harvey IS, Story CR, Knutson D, Whitt-Glover MC. Exploring the Relationship of Religiosity, Religious Support, and Social Support Among African American Women in a Physical Activity Intervention Program. J Relig Health. 2016 Apr;55(2):495-509. doi: 10.1007/s10943-015-0017-6. PMID 25673181
- [Derived] Whitt-Glover MC, Goldmon MV, Karanja N, Heil DP, Gizlice Z. Learning and Developing Individual Exercise Skills (L.A.D.I.E.S.) for a better life: a physical activity intervention for black women. Contemp Clin Trials. 2012 Nov;33(6):1159-71. doi: 10.1016/j.cct.2012.08.003. Epub 2012 Aug 11. PMID 22917598